CLINICAL TRIAL: NCT01732614
Title: Safety Assessment and Therapeutic Effect of Non-damaging Patterned Scanning Laser Phototherapy in Patients With Diffuse Diabetic Macular Edema
Brief Title: Topcon Endpoint Management
Acronym: Topcon EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retinal Consultants of Arizona (Other)
Collaborators: Topcon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Topcon Endpoint Management
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; DME; Laser; Topcon; EndPoint Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topcon Endpoint Management Laser (Experimental)
  Interventions: Procedure: Topcon Endpoint Management laser

INTERVENTIONS:
Procedure: Topcon Endpoint Management laser

SUMMARY:
This trial seeks to prove that sub-lethal laser power levels are as effective and less damaging than traditional laser. Diabetic macular edema (DME) affects approximately 29% of diabetic patients with a disease duration of 20 or more years and is one of the most frequent causes of vision loss in this population. The Early Treatment Diabetic Retinopathy Study (ETDRS) demonstrated a significant benefit of laser photocoagulation for the treatment of clinically significant macular edema, reducing the incidence of vision loss by approximately 50% at 3 years' follow-up.

DETAILED DESCRIPTION:
Sub-visible, non-damaging visible laser (532 nm) exposures of 100 ms in duration resulted in enhanced expression of heat shock proteins in the retina. To test clinical efficacy of sub-visible retinal therapy using ms-range exposures of visible lasers one needs first to establish proper titration methods necessary to assure on one hand the lack of tissue damage, and on the other hand sufficient hyperthermia to elicit cellular response.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have macular edema involving the center of the macula with a corresponding leakage on fluorescein angiography.
* Thickening of the fovea of at least 300 microns (thickness of the central point in OCT) with a standard deviation of the center point <10% and signal strength of ≥ 5 OCT ILM and borders (internal limiting membrane) and RPE (retinal pigment epithelium) properly identified. Also, the initial OCT must be confirmed by repeated measurements on the same day, with the thickness of the central point being within 10% between measurements. In cases where the OCT imaging program can not properly define the limits of ILM and RPE, if the investigator can obtain an estimate of the thickness of the manual by OCT central point of at least 300 microns, the patient will be considered eligible.
* The distance visual acuity in the better eye corrected the study must have an index between 70 and 35 letters inclusive (Snellen equivalent of 20/40 to 20/200).
* Clear media and eye pupil dilation adequate to allow fundus photography with good quality.
* Intraocular pressure not exceeding 21 mmHg.
* The ophthalmologist should feel comfortable with the delay of the focal laser treatment (direct and grid, as needed) by at least 12 weeks in the study eye.
* Patients with diabetes Type I or Type II as defined by WHO criteria of any gender and age ≥ 18 years.
* Ability to provide a written consent.
* Ability to return for all study visits.

Exclusion Criteria:

* Eyes with scatter photocoagulation (PRP) one month prior the enrollment, or eyes where scatter photocoagulation is required now, or it likely to be needed over the next 6months (for example, eyes with high risk PDR DRS not properly treated with photocoagulation).
* Presence of any abnormality that is likely to confound the assessment of the improvement in visual acuity in eyes with macular edema to resolve or improve as an area of hard exudates involving the foveal avascular zone (FAZ - involving 2 or more quadrants centered around the foveal avascular zone), epiretinal membrane associated with signs of contraction and / or significant opacification (ie, striations within the diameter of a disc from the center of the fovea), or the presence of chorioretinal atrophy involving the center of the macula.
* Vitreomacular traction determined clinically and / or OCT, which in the opinion of the investigator, contributes to macular edema (associated or cause a detachment of the fovea) and prevents the improvement with treatment.
* Any cause of macular edema other than DME.
* Atrophy / scar / fibrosis involving the center of the macula, including evidence of atrophy treated with laser within 200 microns of the FAZ.
* Patients who received panphotocoagulation, YAG laser, or peripheral retinal cryoablation (for retinal tears) or focal or grid photocoagulation within the last 12 weeks or more of treatment with focal or grid laser.
* Significant opacities of the optical medium, including cataracts, which may interfere with visual acuity, assessment of toxicity or photography background. Patients will not be included if they have high probability of requiring cataract surgery within the next year.
* Any intraocular surgery within 6 months prior to study entry.
* Prior peeling of epiretinal membrane or inner limiting membrane.
* Any major surgical procedure within one month of study entry
* Prior irradiation of the head region of the eye under study.
* Any previous pharmacological treatment for DME (including corticosteroid intravitreal, subconjunctival or subtenon) or at any time during the last 90 days for any other condition.
* Important known allergies to sodium fluorescein dye used in angiography.
* Acute ocular or periocular infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Visual acuity | 12 months
  Improvement in visual acuity > 10 letters or two lines in the ETDRS chart
Reduction of the central macular thickness by SD-OCT | 12 months
  Reduction of the central macular thickness by SD-OCT

SECONDARY OUTCOMES:
Cessation of leakage areas on FA | 12 months
  Use of fluorescein angiography to assess leakage and identify laser burn

CONTACTS AND LOCATIONS:
Overall Officials: Pravin U Dugel, MD, Principal Investigator — Retinal Consultants of Arizona
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States